CLINICAL TRIAL: NCT04996745
Title: Taking POSNA's OrthoKids to the People: Overcoming Knowledge Disparities in Pediatric Orthopaedic Trauma
Brief Title: Taking POSNA's OrthoKids to the People
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Submitted in error
Sponsor: Louisiana State University Health Sciences Center in New Orleans (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: POSNA's OrthoKids
Record Dates: First submitted 2021-07-27; First posted 2021-08-09 (Actual); Last update posted 2024-08-26 (Actual); Status verified 2024-08

CONDITIONS: Fracture Forearm; Pediatric ALL
Keywords: health literacy; pediatric fractures; OrthoKids
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Patients randomized to the intervention group of the RCT will be given tablet-based education. The first clinic follow-up visit will consist of screening for consent, providing a QR code for Orthokids, and conducting the pre-intervention questionnaire. The pre-intervention questionnaire has two sections with questions pertaining to demographics and orthopedic knowledge. The second clinic follow-up visit will be provided with the tablet for repeat education, with Orthokids and the post-intervention questionnaire will be distributed. The post-intervention questionnaire has two sections with questions pertaining to orthopedic knowledge and satisfaction with care.
  Interventions: Behavioral: Tablet-based educational intervention
- Control Group (No Intervention): Patients randomized to the control group of the RCT will receive the standard clinic experience. This group will not be exposed to any education enrichment about their child's fracture except for the physician's explanation within the exam room.
  The first clinic follow-up visit will consist of screening for consent and conducting the pre-intervention questionnaire. The pre-intervention questionnaire has two sections with questions pertaining to demographics and orthopedic knowledge. The second clinic follow-up visit will consist of conducting the post-intervention questionnaire. The post-intervention questionnaire has two sections with questions pertaining to orthopedic knowledge and satisfaction with care.

INTERVENTIONS:
Behavioral: Tablet-based educational intervention — POSNA's Orthokids website and the article on pediatric forearm fracture will be provided on a tablet. The article provided has two separate tabs, labeled "Condition" and "FAQs", that caregivers will be able to read through. Those who speak Spanish will have the Spanish translated version of Orthokids.
  Arms: Intervention Group

SUMMARY:
The objective of this project is to determine the efficacy of a tablet-based educational intervention at improving orthopaedic health literacy amongst families of pediatric patients treated for fractures in an outpatient setting.

DETAILED DESCRIPTION:
This project aims to reduce knowledge disparity amongst caregivers of patients presenting for pediatric fracture care. At our institution, many patients presenting with fractures do not have easy access to either technology or the internet, preventing caregivers from benefiting from educational tools such as POSNA's OrthoKids®. We are planning to increase access and improve health literacy through a simple intervention of providing tablet-based access to POSNA's Orthokids while families are waiting for their physician. Families will be randomized to either standard waiting room experience vs. tablet-based educational intervention to limit selection bias. A brief pre-visit questionnaire will be completed by all caregivers to assess fracture and cast care knowledge as well as the highest educational degree obtained by the caregiver.

ELIGIBILITY:
Inclusion Criteria (RCT and observational arms):

* Children with forearm fractures who presented to the CHNOLA ED. "Children" are defined as persons under the age of 18 years for this study. "Forearm fracture" is defined as a radial and or ulnar shaft fracture for this study.
* Documented radiographs must show an injury in which the fracture line is wholly located within the diaphysis of the radius or ulna.

Exclusion Criteria (RCT and observational arms):

* Fractures that require internal or external fixation
* Fractures associated with multi-system trauma
* Caregivers that do not speak English or Spanish as their first language

Ages: 0 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2021-10 (Estimated); Primary Completion 2022-08 (Estimated); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
Change in Knowledge questionnaire scores | up to the second clinic followup visit (Average 6 weeks)

SECONDARY OUTCOMES:
Change in caregiver satisfaction scores | up to the second clinic followup visit (Average 6 weeks)
Feedback about the OrthoKids website | up to the second clinic followup visit (Average 6 weeks)

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Hospital of New Orleans, New Orleans, Louisiana, United States